CLINICAL TRIAL: NCT05178589
Title: The Role of Transcutaneous Electrical Nerve Stimulation (TENS) for Menstrual Pain Relief: A Randomized Control Trial
Brief Title: The Role of Transcutaneous Electrical Nerve Stimulation (TENS) for Menstrual Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Associate Professor of Clinical Physical Therapy, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-21-00629
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: This is a randomized cross-over design over the course of 3 menstrual cycles. Each menstruation phase begins on the first day of menstruation until the last day of menstruation (disappearance of bleeding). Each participant will participate in 3 randomized conditions: control (no TENS), one-unit TENS, and two-unit TENS.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control (No Intervention): During the control condition cycle (no TENS), participants will refrain from using or taking other analgesics, besides ibuprofen.
- One Unit TENS (Experimental): Participants will use one-unit TENS set-up where the TENS unit has 2 channels.
  Interventions: Device: One Unit TENS
- Two Unit TENS (Experimental): Participants will use a two-unit TENS set-up where the TENS unit has 4 channels.
  Interventions: Device: Two Unit TENS

INTERVENTIONS:
Device: One Unit TENS — TENS was administered by the participant at home. Application was limited to the abdominal area and instructed to be placed at the location of pain. Single unit TENS was administered via 2 channels. Participants chose an intensity of comfort and continued the treatment for 30-90 minutes per session with unlimited sessions allowed per day.
  Other Names: PowerDot
  Arms: One Unit TENS
Device: Two Unit TENS — TENS was administered by the participant at home. Application was limited to the abdominal area and instructed to be placed at the location of pain. Double unit TENS was administered via 4 channels. Participants chose an intensity of comfort and continued the treatment for 30-90 minutes per session with unlimited sessions allowed per day.
  Other Names: PowerDot
  Arms: Two Unit TENS

SUMMARY:
The present study aims to verify the analgesic potential of a transcutaneous electrical nerve stimulation (TENS) device using patients with primary dysmenorrhea and compare it with a control period without usage.

ELIGIBILITY:
Inclusion Criteria:

* History of lower abdominal pain (dysmenorrhea) for more than 6 consecutive menstrual cycles with a moderate or severe pain rating ≥5 out of 10 over course of last year
* BMI of 18.5-29.9 as a BMI below or above these cut points results in highly varied menstrual cycle lengths
* Not taking contraception or other types of medication that could influence reproductive status
* Regular menstruation
* Medically free from chronic diseases
* Free from known gynecological problems (ie. Endometriosis, Fibroids, Ovarian Cysts)
* History of analgesic pill intake during menstruation
* No pelvic pathology

Exclusion Criteria:

* Amenorrhea
* On a form of contraception
* Secondary dysmenorrhea and/or other gynecological problems that may cause pain
* No discomfort, pain, or other symptoms during menstruation
* History of surgery over lower abdomen area
* Allergy to ibuprofen
* Cardiac disability
* Pacemaker
* Arterial disease
* Uncontrolled hemorrhage
* Blood clots
* Pregnancy or trying to become pregnant
* Cancerous lesions
* Exposed metal implants
* History of seizures
* Sensory or mental impairment
* Unstable fractures

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All menstruating persons are able to participate.
Enrollment: 44 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Analgesic effects of TENS on primary dysmenorrhea. | 1 month
  To determine whether TENS will reduce pain symptoms in those with primary dysmenorrhea. Subjective pain will be assessed using an 11 point visual analog scale (VAS). The scale ranges from 0 to 10, with 0 being no pain and 10 being maximum pain.

SECONDARY OUTCOMES:
Change in analgesic pill consumption during menstruation | 1 month
  Participants will be administered a daily survey where they will be asked to record analgesic pill intake throughout the day.

OTHER OUTCOMES:
The surface area of TENS pain relief | 1 month
  Participants will use either one or 2 unit TENS.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schroeder, PhD, Principal Investigator — Associated Professor
Locations (1):
- University of Southern California Health Sciences Campus Center for Health Professions, Los Angeles, California, United States

REFERENCES:
- [Derived] McLagan B, Dexheimer J, Strock N, Goldstein S, Guzman S, Erceg D, Schroeder ET. The role of transcutaneous electrical nerve stimulation for menstrual pain relief: A randomized control trial. Womens Health (Lond). 2024 Jan-Dec;20:17455057241266455. doi: 10.1177/17455057241266455. PMID 39066557